CLINICAL TRIAL: NCT05221151
Title: Efficacy of Preoperative Melatonin Versus Pregabalin on Intraoperative Anxiolysis and Sedation During Hip Arthroplasty Under Regional Anesthesia
Brief Title: Melatonin vs Pregabalin for Anxiolysis and Sedation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Menoufia University (Other)
Responsible Party: Principal Investigator, mostafa saieed fahim mansour, lecturer, Menoufia University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 1/2022ANET3-B
Record Dates: First submitted 2022-01-07; First posted 2022-02-02 (Actual); Last update posted 2022-12-21 (Actual); Status verified 2022-12

CONDITIONS: Anxiety
Keywords: melatonin; pregabalin
MeSH Terms: conditions — Anxiety Disorders | interventions — Melatonin; Pregabalin; Ondansetron

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- melatonin (Active Comparator): 26 patients will receive melatonin 10 mg
  Interventions: Drug: Melatonin; Drug: Ondansetron 4 MG
- pregabalin (Active Comparator): 26 patients will receive pregabalin 150 mg
  Interventions: Drug: Pregabalin; Drug: Ondansetron 4 MG
- melatonin and pregabalin (Active Comparator): 26 patients will receive melatonin 5 mg plus pregabalin 75 mg
  Interventions: Drug: Melatonin; Drug: Pregabalin; Drug: Ondansetron 4 MG

INTERVENTIONS:
Drug: Melatonin — In the night before surgery, 90 minutes before administering the intrathecal anesthesia and 12 hr after surgery
  Arms: melatonin; melatonin and pregabalin
Drug: Pregabalin — In the night before surgery, 90 minutes before administering the intrathecal anesthesia and 12 hr after surgery
  Arms: melatonin and pregabalin; pregabalin
Drug: Ondansetron 4 MG — before spinal anaesthesia

SUMMARY:
preoperative melatonin, pregabalin or both will be given to all patients preoperative

DETAILED DESCRIPTION:
On arrival at the operating room, continuous electrocardiogram, non-invasive blood pressure and pulse oximetry monitors will be applied. Sedation score (ramsay sedation score)(10) will be recorded on arrival to OR An 18-gauge cannula will be inserted in a peripheral vein and a warmed (37°C) lactated Ringer solution infusion was started. Ondansetron 4 mg will be administered intravenously as a prophylaxis against nausea and vomiting. Thereafter the patient will be supported in the sitting position. Intrathecal anaesthetic (room temperature hyperbaric bupivacaine 0.5% (20 mg) + fentanyl 25 μg (0.5 mL) will be given under complete aseptic technique . The patient was returned to the supine position for 15 min then to lateral position with operative side up.

HR and blood pressure will be measured every 2.5 minutes intraoperatively, however, the values will be recorded in the anesthesia chart only every five minutes for 2 hours then every 15 minutes for 3 hours. Durations will be calculated considering the time of spinal injection as time zero.

Hypotension (SAP<100 mmHg or <80% of the baseline measured before spinal anaesthesia) will be treated by ephedrine 6 mg, to be repeated if inadequate response within 2 minutes. If bradycardia (HR≤60 bpm) developed, atropine (0.6 mg) will be given to restore adequate HR (≥60 bpm).

ELIGIBILITY:
Inclusion Criteria:

* ASA I or II
* patients undergoing hip arthroplasty
* patient consent for spinal anaesthesia
* patient alert, concious and good mental condition

Exclusion Criteria:

* Patients with any neurolgical or psychiatric history before the procedure
* Patients with a history of chronic pain
* patients with known allergy to any of this study drugs
* patients have Any contraindication to neuraxial block.

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2022-01-30 (Actual); Primary Completion 2022-05-02 (Actual); Study Completion 2022-10-02 (Actual)

PRIMARY OUTCOMES:
VAS | on arrival to operating room then every 6 hours untill 48 hours
  change of VAS of the patient on a scale from the night before surgery
Ramsey Sedation scale | on arrival to operating room then every 6 hours untill 48 hours
  change of sedation of the patient on a scale from the night before surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, University Hospitals, Shibīn al Kawm, Menoufia, Egypt

IPD SHARING:
Plan to Share IPD: No